CLINICAL TRIAL: NCT00000596
Title: Diffuse Fibrotic Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2002-02

CONDITIONS: Lung Diseases; Pulmonary Fibrosis; Sarcoidosis
MeSH Terms: conditions — Lung Diseases; Pulmonary Fibrosis; Sarcoidosis | interventions — Prednisone; Cyclophosphamide; Dapsone

INTERVENTIONS:
Drug: prednisone
Drug: cyclophosphamide
Drug: dapsone

SUMMARY:
To determine the effects of cyclophosphamide compared with prednisone, dapsone, or high-dose intermittent 'pulse' therapy with methylprednisolone in patients with idiopathic pulmonary fibrosis. Also, to evaluate the use of intermittent, short-term, high-dose intravenous corticosteroids in patients with sarcoidosis. There were actually four separate clinical trials.

DETAILED DESCRIPTION:
BACKGROUND:

The fibrotic lung diseases represent 15 to 20 percent of the non-infectious disorders of the lung. Idiopathic pulmonary fibrosis, one of the 10 general groups of fibrotic lung disorders, is a chronic and devastating illness resulting in death within an average of 4 to 5 years from the onset of symptoms. Although 5 to 10 percent of these patients respond to corticosteroids, there is no known treatment for the remainder.

Sarcoidosis, a generalized disorder characterized by epithelioid cell granuloma formation in affected organs, especially the lung and lymphoid tissue, has a clinical course that varies considerably from patient to patient and, in some cases, resolves spontaneously. In other cases, intermittent pneumonitis develops, which may result in a permanent loss of lung function. Large intermittent doses of corticosteroids might be superior to conventional high-dose corticosteroids in patients with pulmonary sarcoidosis which has not resolved spontaneously.

DESIGN NARRATIVE:

In the randomized, non-blind cyclophosphamide versus prednisone trial, 25 to 50 patients with idiopathic pulmonary fibrosis were assigned to treatment with prednisone or cyclophosphamide. At the end of 52 weeks of drug therapy, both groups were treated using conventional medical therapies. In the non-randomized dapsone trial, 10 fibrotic patients were treated with dapsone and prednisone for one year. In the double-blind, randomized methylprednisolone trial, 25 to 50 patients were given low-dose methylprednisolone, and, in addition, all patients were randomized to either high-dose methylprednisolone treatment or to placebo at weekly intervals for one year. In the randomized, double-blind, high-dose corticosteroid trial, 25 to 50 patients with pulmonary sarcoidosis were given a short intense course of high-dose methylprednisolone or a placebo for 6 weeks.

The study completion date listed in this record was inferred from the last publication listed in the Citations section of this study record.

ELIGIBILITY:
No eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1978-06; Study Completion 1983-01 (Actual)

REFERENCES:
- [Background] Keogh BA, Bernardo J, Hunninghake GW, Line BR, Price DL, Crystal RG. Effect of intermittent high dose parenteral corticosteroids on the alveolitis of idiopathic pulmonary fibrosis. Am Rev Respir Dis. 1983 Jan;127(1):18-22. doi: 10.1164/arrd.1983.127.1.18. PMID 6849542